CLINICAL TRIAL: NCT05445505
Title: Neuroprotective Effects of Intermittent Theta Burst Stimulation in Parkinson's Disease: a Delayed-start Randomized Double-blind Sham Controlled Study
Brief Title: Neuroprotective Effects of iTBS in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022043
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-05

CONDITIONS: Neuroprotection; Parkinson Disease; Intermittent Theta Burst Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early-start single iTBS group (Active Comparator): The intensive period: 2 weeks The maintenance period: 12 weeks
  Interventions: Device: intermittent theta burst stimulation
- Early-start double iTBS group (Active Comparator): The intensive period: 2 weeks The maintenance period: 12 weeks
  Interventions: Device: intermittent theta burst stimulation
- Delayed-start single iTBS group (Sham Comparator): The intensive period: sham/iTBS, 2 weeks The maintenance period: daily sham/iTBS, 12 weeks
  Interventions: Device: intermittent theta burst stimulation; Device: sham iTBS
- Delayed-start double iTBS group (Sham Comparator): The intensive period: sham/iTBS, 2 weeks The maintenance period: twice daily sham/iTBS, 12 weeks
  Interventions: Device: intermittent theta burst stimulation; Device: sham iTBS

INTERVENTIONS:
Device: intermittent theta burst stimulation — iTBS is a new form of excitatory rTMS treatment that is less time-consuming and more effective than traditional rTMS in a single treatment session.
  Other Names: iTBS
Device: sham iTBS — The pseudo-stimulation device looks and sounds the same as the iTBS device
  Arms: Delayed-start double iTBS group; Delayed-start single iTBS group

SUMMARY:
Intermittent theta burst stimulation (iTBS) is an emerging non-invasive neuron regulation technique, which is widely used in neuropsychiatry for a variety of diseases and is widely accepted by patients due to its non-invasive, operable and relatively precise localization. Combining the results of previous studies and our group's previous research, sixty qualified PD patients would be enrolled to conduct a prospective single-center randomized double-blind sham controlled clinical trial to verify the long-term curative effects of iTBS treatment protocol and explore the neuron-protection of iTBS on neuronal loss of PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet the revised clinical diagnostic criteria for Parkinson's disease of the Movement Disorder Society (MDS) International (2015 version).
* aged >20 years and <80 years, regardless of gender.
* 2 ≤ Hoehn-Yahr stage≤ 4.
* Maintain medication stability during the study period.
* Good compliance, written informed consent, and consent for long-term interventional treatment with iTBS.

Exclusion Criteria:

* Patients with severe neuropsychiatric disorders or previous history of severe neurological disorders (e.g., epilepsy, cerebrovascular accidents, etc.) or history of traumatic brain injury or brain surgery.
* Patients with significant cognitive impairment (MMSE < 24) or inability to complete questionnaires independently.
* Prior treatment with TMS, DBS or SCS.
* Severe physical illness and any physical illness that can precipitate epilepsy or intracranial hypertension, including cardiovascular and respiratory disease.
* Have human implantable materials such as intracranial stents, pacemakers, coronary stents, cochlear implants, etc.
* Are currently taking other investigational drugs.
* Any other condition that the investigator deems unsuitable for participation in this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Group differences of part 3 of Unified Parkinson Disease Rating Scale (UPDRS) changes | 28 weeks
  Compare the changes in UPDRS scores from baseline to post-iTBS in the four intervention groups (UPDRS part3: range 0~72, higher score is related to a worse outcome).

SECONDARY OUTCOMES:
Group differences of Hoehn-Yahr stage | 28 weeks
  Compare the changes in Hoehn-Yahr stage from baseline to post-iTBS in the four intervention groups (H-Y stage: range 0~5, higher score is related to a worse outcome).
Group differences of Berg Balance Scale (BBS) changes | 28 weeks
  Compare the changes in BBS scores from baseline to post-iTBS in the four intervention groups (BBS: range 0~56, higher score is related to a better outcome).
Group differences of Hamilton depression scale-17 (HAMD-17) changes | 28 weeks
  Compare the changes in HAMD-17 scores from baseline to post-iTBS in the four intervention groups (HAMD-17: range 0~38, higher score is related to a worse outcome).
Group differences of Hamilton Anxiety Scale (HAMA) changes | 28 weeks
  Compare the changes in HAMA scores from baseline to post-iTBS in the four intervention groups (HAMA: range 0~64, higher score is related to a worse outcome).
Group differences of Mini-mental State Examination (MMSE) changes | 28 weeks
  Compare the changes in MMSE scores from baseline to post-iTBS in the four intervention groups (MMSE: range 0~30, higher score is related to a better outcome).
Group differences of Montreal Cognitive Assessment (MoCA) changes | 28 weeks
  Compare the changes in MoCA scores from baseline to post-iTBS in the four intervention groups (MoCA: range 0~30, higher score is related to a better outcome).
Group differences of 39-item Parkinson's Disease Questionnaire (PDQ-39) changes | 28 weeks
  Compare the changes in PDQ-39 scores from baseline to post-iTBS in the four intervention groups (PDQ-39: range 0~156, higher score is related to a worse outcome).
Group differences of 16-item Sniffin' Sticks test (SS-16) changes | 28 weeks
  Compare the changes in SS-16 scores from baseline to post-iTBS in the four intervention groups (SS-16: range 0~16, higher score is related to a better outcome).
Group differences of Wexner changes | 28 weeks
  Compare the changes in Wexner scores from baseline to post-iTBS in the four intervention groups (Wexner: range 0~30, higher score is related to a worse outcome).
Group differences of adverse event | 28 weeks
  Compare the adverse event in four intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, Professor, Study Chair — Department of Neurology, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) was available to other researchers.